CLINICAL TRIAL: NCT00619931
Title: A Multiple-Dose Study to Assess the Safety, Tolerability, and Steady State Pharmacokinetics of APD791 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APD791-002
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Healthy adult volunteers
MeSH Terms: interventions — APD791

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): APD791 or placebo
  Interventions: Drug: APD791
- 2 (Experimental): APD791 or placebo
  Interventions: Drug: APD791
- 3 (Experimental): APD791 or placebo
  Interventions: Drug: APD791
- 4 (Experimental): APD791 or placebo
  Interventions: Drug: APD791
- 5 (Experimental): APD791 or placebo
  Interventions: Drug: APD791

INTERVENTIONS:
Drug: APD791 — APD791 or matching placebo in escalating doses

SUMMARY:
The APD791-002 study is designed primarily to evaluate the safety, tolerability, and pharmacokinetics of APD791 when administered for 7 days to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women, ages 19-45
* Non smokers

Exclusion Criteria:

* History of a bleeding disorder
* Use of any drug known to have an effect on coagulation or clotting or any anti-platelet therapy within 2 weeks of the screening
* Recently donated blood or had significant blood loss
* Current use of a prescription medication
* Pregnant females

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety measures to include adverse events, vital signs, 12-lead ECGs, physical examinations, and clinical lab parameters | Throughout study duration

SECONDARY OUTCOMES:
Pharmacokinetic assessments | Throughout study duration
Pharmacodynamic assessments (e.g., platelet function) | Throughout study duration

CONTACTS AND LOCATIONS:
Overall Officials: James Kisicki, MD, Principal Investigator — MDS Pharma Services; Christen M Anderson, MD, PhD, Study Director — Arena Pharmaceuticals
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States

REFERENCES:
- See also: Arena Home Page — http://www.arenapharm.com